CLINICAL TRIAL: NCT06522425
Title: Evaluation of the Usability of Mindfulness-based Serious Games for Pediatric Patient Who Need Pain Control
Brief Title: Usability Evaluation of a Mindfulness-based Serious Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-08-073
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic
Keywords: Pain Management, Mindfulness, Serious Game
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- professionals (Experimental): This arm includes 9 professionals (including medical staff, child development specialists, and psychologists). All participants will use the mindfulness-based serious game designed for pain management and will complete usability surveys and participate in interviews to provide feedback on their experience.
  Interventions: Other: mindfulness-based serious games
- Users(pediatric patients) (Experimental): This arm includes 10 users (pediatric patients aged 5-17 years who are taking adjuvant analgesics or narcotic/non-narcotic analgesics for pain control). All participants will use the mindfulness-based serious game designed for pain management and will complete usability surveys and participate in interviews to provide feedback on their experience.
  Interventions: Other: mindfulness-based serious games

INTERVENTIONS:
Other: mindfulness-based serious games — The intervention consists of a single session using a digital serious game designed to teach mindfulness techniques for pain management. In addition to explaining mindfulness concepts, the game provides a variety of mindfulness exercises to help users manage and reduce pain perception. For example, it involves relaxation through breathing or becoming aware of the state of one's body and mind. Additionally, it includes various interaction elements such as touch, voice, and motion controls to increase user immersion.

SUMMARY:
The purpose of this study is to evaluate the usability of a mindfulness-based serious game developed for pediatric and adolescent patients who require pain management during their disease treatment. We conducted usability evaluations targeting both professional and user groups. Both groups experienced the mindfulness-based serious game and then participated in a usability survey and interview.

DETAILED DESCRIPTION:
Background : Pain management is a critical aspect of treatment for pediatric and adolescent patients, especially those undergoing long-term or chronic disease management. Traditional pain management strategies often include pharmacological interventions, which may not be sufficient on their own and can have undesirable side effects. Consequently, there is a growing interest in complementary approaches that can enhance pain management and provide holistic care.

Mindfulness-based interventions have been shown to be effective in managing chronic pain by helping individuals develop a greater awareness of their physical and emotional states, thereby reducing the perception of pain. Serious games, which incorporate elements of play and interaction, offer a novel and engaging way to deliver mindfulness training. These games can be particularly appealing to younger patients, making it easier to integrate mindfulness practices into their daily routines.

Objective : The purpose of this study was to evaluate the usability of a mindfulness-based serious game developed for pediatric and adolescent patients who require pain management during their disease treatment.

Design: mixed-methods design Setting: In the emergency department at Samsung Medical Center Enrollment : 9 professionals (e.g., medical staff, child development specialists, and psychologists) and 10 pediatric and adolescent patients.

Intervention : Both professional and pediatric and adolescent patient groups experience a mindfulness-based functional game developed for pain management through a tablet.

Scoring : Usability is measured using the MARS (Mobile Application Rating Scale) and uMARS (user version of the Mobile Application Rating Scale) in a group of professionals and pediatric and adolescent patients. (Full score of MARS: 145, Full score of uMARS: 130).

Study period : For 1 hour after study enrollment, Usability survey : After experiencing a mindfulness-based functional game

ELIGIBILITY:
1. Users(Pediatric Patients)

   * Inclusion Criteria:

     1. Pediatric patients aged 5-17 years.
     2. Currently taking adjuvant analgesics or narcotic/non-narcotic analgesics for pain control.
     3. Able to provide voluntary assent and have parental/guardian consent.
   * Exclusion Criteria:

     1. Diagnosed with a psychiatric disorder characterized by psychotic features.
     2. Have visual or auditory impairments that would make it difficult to understand and play the game.
2. Professionals

   * Inclusion Criteria:

     1. Medical staff specializing in pediatric care or individuals with a doctoral degree in child development or psychology
     2. Able to provide voluntary informed consent.
   * Exclusion Criteria:

     1. Have visual or auditory impairments that would make it difficult to understand and play the game.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Usability Evaluation of the Mindfulness-Based Serious Game | Immediately post-intervention
  The usability of the mindfulness-based serious game will be measured using the Mobile Application Rating Scale (MARS) and its user version (uMARS). These scales assess the app's engagement, functionality, aesthetics, information, subjective quality and app-specific quality.

SECONDARY OUTCOMES:
Qualitative Feedback from Interviews | Immediately post-intervention
  Qualitative feedback will be collected through interviews conducted immediately after the intervention. These interviews will gather detailed insights into participants' experiences, including the game's usability, perceived benefits, ease of use, and overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Meong hi Son, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Centre, Seoul, South Korea